CLINICAL TRIAL: NCT01034761
Title: Using Clinical Alerts in a Computerized Provider Order Entry System to Decrease Inappropriate Medication Prescribing Among Hospitalized Elders
Brief Title: Using Clinical Alerts to Decrease Inappropriate Medication Prescribing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Linda Canty, MD, Assistant Clinical Professor of Medine, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 132454
Record Dates: First submitted 2009-12-15; First posted 2009-12-17 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Elderly
Keywords: Electronic prescribing; Inappropriate medications; Patient safety; Elderly patients in the hospital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pop-up alerts (Experimental): Providers will receive pop-up alerts in the electronic medical record when prescribing one of the specified medications from the Beers list.
  Interventions: Behavioral: Pop-up alert
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Pop-up alert — Pop-up alert in the electronic medical record whenever the provider enters an order for a specified high risk medication from the Beers list.
  Arms: Pop-up alerts

SUMMARY:
Introduction:

The Beers list identifies medications that should be avoided in persons 65 years or older because they are ineffective, pose an unnecessarily high risk, or a safer alternative is available. In a recent study, we found a high rate of prescribing of Beers list medications to hospitalized patients. At Baystate, 41% of medical patients received at least one Beers list drug classified as "high severity," meaning it carried a high risk for an adverse drug reaction, while 5% received 3 or more. Some Beers drugs have been associated with delirium and falls. When compared to Baystate patients who did not receive a high severity medication, those who did had an increased risk of mortality (7.8% vs. 5.2%), longer length of stay (5.5 days vs. 3.9 days) and higher costs ($11,240 vs. 6243).

Specific Aims:

1. Quantify the impact of synchronous electronic alerts on physician prescribing of high-severity Beers' list drugs to hospitalized patients over the age of 65 years.
2. Compare physician reactions to each drug-specific alert

Project Description:

We will develop a series of clinical alerts in CIS, Baystate's computerized provider order entry system, to reduce the use of potentially inappropriate medications among hospitalized elders. We will randomize providers to electronic alerts or usual care. Whenever a provider randomized to alerts attempts to place an order for a high-risk medication on the Beers list and the intended recipient is over 65 years of age, a synchronous alert (i.e. a "pop-up") will inform the physician about the risks associated with the medication and will propose safer alternatives.

We will collect data on physician ordering and patient outcomes comparing the number of Beers list prescriptions from providers receiving electronic alerts to those not receiving alerts. Our anticipated outcome is a decrease in inappropriate prescribing during the period when the electronic alerts are activated. Other potential outcomes include decrease in length of stay and a decrease in falls.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with Age > 65

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 719 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The percentage of elderly patients who receive a specified high-risk medication from the Beer's list. | Earlier of hospital stay or end of study

SECONDARY OUTCOMES:
The average number of specified high risk medications prescribed per patient. | Earlier of hospital stay or end of study
Restraint use | Earlier of hospital stay or end of study
Falls | Earlier of hospital stay or end of study
Length of stay | Earlier of hospital stay or end of study
Total Cost | Earlier of hospital stay or end of study
Discharge status | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Canty, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

REFERENCES:
- [Derived] Cole JA, Goncalves-Bradley DC, Alqahtani M, Barry HE, Cadogan C, Rankin A, Patterson SM, Kerse N, Cardwell CR, Ryan C, Hughes C. Interventions to improve the appropriate use of polypharmacy for older people. Cochrane Database Syst Rev. 2023 Oct 11;10(10):CD008165. doi: 10.1002/14651858.CD008165.pub5. PMID 37818791